CLINICAL TRIAL: NCT03495050
Title: BIVOLUTX: Bicuspid Aortic Stenosis With Evolut Platform International Experience.
Acronym: BIVOLUTX
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Clinique Pasteur (Other)
Responsible Party: Principal Investigator, Didier TCHETCHE, Head of structural heart disease program, Clinique Pasteur
Other Study IDs: 2018-A00290-55
Record Dates: First submitted 2018-03-03; First posted 2018-04-11 (Actual); Last update posted 2018-06-12 (Actual); Status verified 2018-06

CONDITIONS: Bicuspid Aortic Valve
Keywords: Bicuspid; TAVI; TAVR; self-expanding; Evolut
MeSH Terms: conditions — Bicuspid Aortic Valve Disease | interventions — Transcatheter Aortic Valve Replacement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: Transcatheter Aortic Valve Implantation — Transcatheter treatment of bicuspid aortic stenosis with the Evolut Pro/XL platform
  Other Names: Transcatheter Aortic Valve Replacement

SUMMARY:
Prospective non interventional, observational registry of 150 patients undergoing TAVI with Evolut platform for bicuspid aortic stenosis.

DETAILED DESCRIPTION:
Study Design Study Design: prospective non-interventional multicenter registry Screening: MSCT submitted to core lab & sizing strategy pre-declared (annular sizing, supra-annular sizing, mix of both methods) Follow up: MSCT and TTE to cooper lab

TAVI treatment Predilatation according to aortic annulus Dmin Evolut Pro (23-26-29) and Evolut R 34 XL Annular anchoring of the THV Postdilatation according to the operators' discretion Study Population All consecutive patients presenting with severe and symptomatic bicuspid aortic valve stenosis or mixed disease

Inclusion Criteria 1. Age ≥18 years. 2. NYHA≥2 and/or syncope and/or angina. 3. Patient judged by the Heart Team as indicated for TAVI. 4. Anatomical suitability for transfemoral-TAVI with Evolut Pro or Evolut R XL, based on MSCT assessment.

5. Estimated life-expectancy>1 year.

Exclusion Criteria 1. Age <18 years 2. Asymptomatic patients 3. Estimated life expectancy<1 year 4. Pure aortic regurgitation. 5. LVEF<20% 6. No baseline MSCT evaluation. 7. Unsuitable aortic root anatomy for Evolut Pro or XL. 8. Unsuitable peripheral vasculature for transfemoral Evolut Pro or XL. Primary Endpoint Valve performane Secondary endpoints 30 day and 1 year mortality Patient-prosthesis mismatch Ellipticity index at 30 days Follow-up 30 days: physical examination, ECG, TTE /MSCT upon operators' judgement

1 year: physical examination, ECG, TTE.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years.
2. NYHA≥2 and/or syncope and/or angina.
3. Patient judged by the Heart Team as indicated for TAVI.
4. Anatomical suitability for transfemoral-TAVI with Evolut Pro or Evolut R XL, based on MSCT assessment.
5. Estimated life-expectancy>1 year.

Exclusion Criteria:

1. Age <18 years
2. Asymptomatic patients
3. Estimated life expectancy<1 year
4. Pure aortic regurgitation.
5. LVEF<20%
6. No baseline MSCT evaluation.
7. Unsuitable aortic root anatomy for Evolut Pro or XL.
8. Unsuitable peripheral vasculature for transfemoral Evolut Pro or XL.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All consecutive patients presenting with severe and symptomatic bicuspid aortic valve stenosis or mixed disease
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2018-02-21 (Actual); Primary Completion 2019-05 (Estimated); Study Completion 2020-05 (Estimated)

PRIMARY OUTCOMES:
Valve performance | 30 days
  effective orifice area<0.85 cm2/m2 and/or mean gradient>20 mmHg and/or aortic regurgitation>moderate
Valve performance | one year
  effective orifice area<0.85 cm2/m2 and/or mean gradient>20 mmHg and/or aortic regurgitation>moderate

SECONDARY OUTCOMES:
mortality | 30 days and one year
Patient-prosthesis mismatch | 30 days and 1 year
  indexed effective area <0.65 cm2/m2
Ellipticity index at 30 days | 30 days

CONTACTS AND LOCATIONS:
Locations (1):
- Clinique Pasteur, Toulouse, Occitanie, France

IPD SHARING:
Plan to Share IPD: Undecided
Mutual ananymized database. Substudies anticipated.

REFERENCES:
- [Derived] Tchetche D, de Biase C, van Gils L, Parma R, Ochala A, Lefevre T, Hovasse T, De Backer O, Sondergaard L, Bleiziffer S, Lange R, Kornowski R, Landes U, Norgaard BL, Biasco L, Philippart R, Molina-Martin de Nicolas J, Mylotte D, Lemee C, Dumonteil N, Van Mieghem NM. Bicuspid Aortic Valve Anatomy and Relationship With Devices: The BAVARD Multicenter Registry. Circ Cardiovasc Interv. 2019 Jan;12(1):e007107. doi: 10.1161/CIRCINTERVENTIONS.118.007107. PMID 30626202